CLINICAL TRIAL: NCT02896985
Title: A Cohort Study to Evaluate the Effectiveness of Drug Concentrations in Predicting Recapture of Response With Weekly ADAlimumab in Crohn's Disease Subjects With Secondary Loss of Response (PRADA)
Brief Title: Observational Study Evaluating the Effectiveness of Drug Concentration to Predict the Recapture of Response in Crohn's Disease Patients With Loss of Response ( PRADA )
Acronym: PRADA
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-770
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Crohn's Disease
Keywords: Patient Reported Outcome 2 (PRO 2); C-Reactive Protein (CRP); Adalimumab; Harvey Bradshaw Index (HBI); Therapeutic Drug Monitoring (TDM); Anti-Adalimumab Antibody (AAA)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Crohn's disease: Participants who have developed LOR to adalimumab after a minimum of 16 weeks of treatment.

SUMMARY:
This is a multi-center study that explores the relationship between recapture of response with escalation to weekly adalimumab and trough adalimumab concentration before escalation in patients experiencing lack of response (LOR).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Crohn's Disease.
* Treatment with adalimumab, for a minimum of 16 weeks, as per clinical practice, at a dose of 160 mg at week 0, 80 mg at week 2, and then 40 mg q2w with a documented response as defined by the investigator.
* Current evidence of active inflammatory disease/LOR defined as the presence of active inflammation (confirmed with a CRP ≥ 5 mg/L and/or a fecal calprotectin ≥ 250µg/g.
* Ability of subject to participate fully in all aspects of this clinical trial.
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* Primary non-responders to 16 weeks of adalimumab therapy.
* Received any investigational drug within the 16 weeks of adalimumab therapy.
* Serious underlying disease other than CD that, in the opinion of the investigator, may interfere with the subject's ability to participate fully in the study.
* History of alcohol or drug abuse that, in the opinion of the investigator, may interfere with the subject's ability to comply with the study procedures.
* Stools positive for Clostridium difficile.
* Pregnant or lactating women.
* Current enrolment in any other interventional research study.
* Presence of perianal or abdominal abscess.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled from approximately 15 to 20 investigative sites in Canada where such Therapeutic Drug Monitoring/Anti-Adalimumab Antibody (TDM/AAA) testing at the point of patient LOR and pre-dose escalation to Every Week (EW) occurs.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Explore the relationship between drug concentration at baseline and recapture of response | At Week 12
  Logistic regression analysis will be used to model the relationship between drug concentration at baseline and recapture of response.

SECONDARY OUTCOMES:
Explore the relationship between trough adalimumab concentrations at baseline and change in patient reported outcome 2 (PRO2) | From Week 0 to Week 12
  Covariance analysis is used.
Explore the relationship between trough adalimumab concentrations at baseline and change in C-reactive protein (CRP) | From Week 0 to Week 12
  Covariance analysis is used.
Explore the relationship between trough adalimumab concentrations at baseline and change in fecal calprotectin | From Week 0 to Week 12
  Covariance analysis is used.
Proportion of participants requiring steroids or additional therapy | Up to Week 12
  Assessing participants that require steroids or additional therapy
Proportion of participants with 50% drop from screening in CRP or calprotectin | At Week 12
  Assessing participants with 50% drop in CRP or calprotectin.
Explore the relationship between changes in HBI between screening and final trough adalimumab concentrations | At Week 12
  Covariance analysis is used.
Proportion of participants with clinical remission PRO2 < 8 | At Week 12
  PRO2 was developed based on FDA guidance for use of patient reported outcomes.
Proportion of participants with normalization of CRP or fecal calprotectin | At Week 12
  Assessing participants with normalization of CRP (<5mg/dl) or fecal calprotectin (<150ug/ml)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (24):
- Canada (24):
  - University of Calgary /ID# 157893, Calgary, Alberta
  - South Edmonton Gastroenterolog /ID# 170934, Edmonton, Alberta
  - Columbia Gastro Mgmnt Ltd /ID# 152507, New Westminster, British Columbia
  - GIRI Gastrointestinal Research Institute /ID# 201259, Vancouver, British Columbia
  - Discovery Clinical Services /ID# 154682, Victoria, British Columbia
  - Percuro Clinical Research, Ltd /ID# 202502, Victoria, British Columbia
  - Winnipeg Regional Health Autho /ID# 200115, Winnipeg, Manitoba
  - Dr. Everett Chalmers Reg Hosp. /ID# 171560, Fredericton, New Brunswick
  - Qe Ii Hsc /Id# 152454, Halifax, Nova Scotia
  - Dr. Mark Lee Medicine Professi /ID# 153127, Cambridge, Ontario
  - McMaster University Med Cent /ID# 151996, Hamilton, Ontario
  - London Health Sciences Centre /ID# 152508, London, Ontario
  - Jeffrey So Medicine Professional Corporation /ID# 168268, Oakville, Ontario
  - Taunton surgical centre /ID# 151998, Oshawa, Ontario
  - The Ottawa Hospital /ID# 153771, Ottawa, Ontario
  - Mount Sinai Hosp.-Toronto /ID# 155262, Toronto, Ontario
  - Dr O Tarabain Medicine Prof Corp /ID# 163125, Windsor, Ontario
  - CISSS de la Monteregie /ID# 162724, Greenfield Park, Quebec
  - Hopital Hotel-Dieu de Levis /ID# 155493, Lévis, Quebec
  - Hospital Maisonneuve-Rosemont /ID# 155184, Montreal, Quebec
  - McGill Univ HC /ID# 151997, Montreal, Quebec
  - Clinique MEDI-CLE /ID# 153772, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 157976, Sherbrooke, Quebec
  - Royal Uni Saskatchew(CTSU) /ID# 162316, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-770.pdf